CLINICAL TRIAL: NCT01223352
Title: An Open-label, Prospective Multicenter Study to Assess the Pharmacokinetics, Tolerability, Safety and Efficacy of the Pediatric Formulation of Bosentan Two Versus Three Times a Day in Children With Pulmonary Arterial Hypertension
Brief Title: Effects of Two Dosing Regimens of Bosentan in Children With Pulmonary Arterial Hypertension
Acronym: FUTURE 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC-052-373
Record Dates: First submitted 2010-10-12; First posted 2010-10-19 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; children; pediatric; bosentan
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bosentan 2 mg/Kg t.i.d. (Experimental): 2 mg/kg bosentan administered three times a day (morning, afternoon, evening) for a planned duration of 24 weeks
  Interventions: Drug: bosentan
- Bosentan 2 mg/Kg b.i.d. (Experimental): 2 mg/kg bosentan administered twice daily (morning and evening) for a planned duration of 24 weeks
  Interventions: Drug: bosentan

INTERVENTIONS:
Drug: bosentan — 32 mg quadrisected dispersible tablet. The dosage of bosentan (2 mg/Kg) was adjusted according to the patient's body weight at initiation of the study treatment. Dosage readjustment was permitted after 12 weeks of treatment.
  Other Names: Tracleer; ACT-050088

SUMMARY:
The primary objective of AC-052-373 was to assess the pharmacokinetic (PK) profile of two dosing regimens of the pediatric formulation of bosentan in children with pulmonary arterial hypertension (PAH) <12 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. PAH diagnosis confirmed with right heart catheterization (RHC):

   * Idiopathic or heritable PAH, or
   * Associated PAH persisting after complete repair of a congenital heart defect (PAH has to be persistent for at least 6 months after surgery) or
   * PAH-Congenital Heart Disease (PAH-CHD) associated with systemic-to-pulmonary shunts (after global amendment dated 09 May 2012)
2. World Health Organization functional Class (WHO FC) I, II or III
3. Male or female ≥ 3 months and < 12 years of age (maximum age at randomization is 11.5 years)
4. Body weight ≥ 3.5 kg
5. Peripheral oxygen saturation (SpO2) ≥ 88% (at rest, on room air)
6. Baseline PAH-therapy (Calcium channel blocker, bosentan, prostanoid, phosphodiesterase type-5 inhibitor) if present, has to be stable for at least 3 months prior to screening. During the study, all background treatments should remain stable
7. Signed informed consent by the parents or legal representatives

Exclusion Criteria:

1. PAH etiologies other than listed above
2. Non-stable disease status
3. Need or plan to wean patient from intravenous epoprostenol or intravenous or inhaled iloprost
4. Systolic blood pressure < 80% of the lower limit of normal range
5. Aspartate aminotransferase and/or alanine aminotransferase values > 1.5 times the upper limit of normal range.
6. Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C
7. Hemoglobin and/or hematocrit levels < 75% of the lower limit of normal range.
8. Known intolerance or hypersensitivity to bosentan or any of the excipients of the dispersible Tracleer tablet
9. Treatment with forbidden medication within 2 weeks or at least 5 times the half-life prior to randomization, whichever is the longest:

   * Glibenclamide (glyburide)
   * Cyclosporin A
   * Sirolimus
   * Tacrolimus
   * Fluconazole
   * Rifampicin (rifampin)
   * Ritonavir
   * Co-administration of CYP2C9 inhibitors (e.g., amiodarone, voriconazole) and moderate/strong CYP3A4 inhibitors (e.g., amprenavir, erythromycin, ketoconazole, diltiazem, itraconazole)
   * Endothelin receptor antagonists (ERAs) other than bosentan
10. Treatment with another investigational drug within 1 month prior to randomization or planned treatment

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2011-03-08 (Actual); Primary Completion 2013-04-03 (Actual); Study Completion 2013-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andjela Kusic-Pajic, MD, Study Director — Actelion

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-five expert pediatric centers were initiated but only thirty of them enrolled children with pulmonary arterial hypertension (PAH)
Groups:
- Bosentan 2 mg/kg t.i.d.: 2 mg/kg bosentan (dispersible tablets) was administered orally three times a day (t.i.d.) for a planned duration of 24 weeks
- Bosentan 2 mg/kg b.i.d.: 2 mg/kg bosentan (dispersible tablets) was administered orally twice daily (b.i.d.) for a planned duration of 24 weeks
Period: Overall Study
Arm/Group | Bosentan 2 mg/kg t.i.d. | Bosentan 2 mg/kg b.i.d.
Started | 31 | 33
Completed | 31 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bosentan 2 mg/kg t.i.d. | Bosentan 2 mg/kg b.i.d. | Total
Number analyzed (Participants) | 31 | 33 | 64
Age, Continuous [Mean (Standard Deviation); unit: Years] — This is the age reported at the screening visit which had to be performed within 4 weeks prior to randomization
  Years | 5.2 (3.81) | 4.5 (3.35) | 4.8 (3.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 18 | 28
  Male | 21 | 15 | 36
Region of Enrollment [Number; unit: Participants]
  Australia | 2 | 0 | 2
  Belarus | 1 | 2 | 3
  China | 2 | 4 | 6
  Czech Republic | 1 | 1 | 2
  France | 1 | 4 | 5
  Germany | 3 | 1 | 4
  Hungary | 3 | 0 | 3
  India | 1 | 2 | 3
  Israel | 0 | 2 | 2
  Italy | 1 | 0 | 1
  Mexico | 1 | 0 | 1
  Poland | 2 | 3 | 5
  Russia | 4 | 6 | 10
  Serbia | 2 | 3 | 5
  South Africa | 4 | 2 | 6
  Spain | 1 | 2 | 3
  USA | 1 | 1 | 2
  Ukraine | 1 | 0 | 1
Etiology of pulmonary arterial hypertension (PAH) [Count of Participants; unit: Participants] — Children included in the study had a diagnosis of PAH belonging to one of the following categories:
  * Idiopathic PAH
  * Heritable PAH
  * Associated PAH persisting after complete repair of a congenital heart defect
  * PAH-congenital heart disease (PAH-CHD) associated with open shunts
  Participants
    Idiopathic | 15 | 14 | 29
    Heritable | 0 | 2 | 2
    PAH-Congenital heart disease | 2 | 6 | 8
    Associated PAH | 13 | 11 | 24
    Missing data | 1 | 0 | 1
World Health Organization functional class (WHO FC) [Number; unit: Participants] — The World Health Organization (WHO) defines 4 classes to classify the functional status of patients with pulmonary hypertension:
  Class I (FC I): No limitation of physical activity; Class II (FC II): Slight limitation of physical activity; Class IIII (FC III): Marked limitation of physical activity; Class IV (FC IV): Inability to carry out any physical activity without symptoms.
  WHO FC at Day 1, before first study drug administration, are reported as baseline values here.
  Participants
    FC I | 10 | 9 | 19
    FC II | 15 | 12 | 27
    FC III | 6 | 12 | 18
PAH-specific therapy at baseline [Number; unit: Participants] — PAH-specific therapy at Day 1, before first study drug administration, are reported as baseline values here.
  Participants
    Bosentan (adult tablet formulation) | 4 | 3 | 7
    Prostanoid | 1 | 0 | 1
    Phosphodiesterase type-5 (PDE-5) inhibitor | 13 | 10 | 23
    Bosentan / PDE-5 inhibitor combination | 2 | 2 | 4
    Bosentan /PDE-5 inhibitor /Prostanoid combination | 2 | 5 | 7
    None | 9 | 13 | 22

OUTCOME MEASURES:

1. Primary Outcome: Dose-corrected Daily Exposure [AUC(0-24c)] to Bosentan
Description: Daily exposure was measured by the area under the plasma concentration-time curve over a period of 24 hours [AUC(0-24)].
  Concentrations of bosentan were measured directly in blood samples collected prior to study drug administration and up to 8 hours or up to 12 hours post-dose for the t.i.d and b.i.d. dosing regimen, respectively. AUC(0-24) was calculated as a multiple of AUCtau, which is the AUC over a dosing interval (AUCtau x 2 for the b.i.d. dosing regimen and AUCtau x 3 for the t.i.d. regimen). As the smallest dose unit was 8 mg (1/4 tablet), it was not possible to achieve the exact target dose of 2 mg/kg. Therefore, AUC(0-24) was corrected to 2 mg/kg (target dose) [AUC(0-24c)].
Time Frame: 0, 0.5, 1, 3, 5 (or 7.5), 8 (or 12 hours) post-dose at Week 4, after at least 2 weeks of stable study drug treatment
Population: Per-protocol PK analysis set (PK set): All patients included in the bosentan 2 mg/kg b.i.d. and bosentan 2 mg/kg t.i.d. groups who received at least one dose of bosentan and who were able to provide at least 5 blood samples for PK assessments and who did not violate the protocol in a way that might affect the evaluation of the PK main endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Groups:
- Bosentan 2 mg/kg t.i.d. (PK Set): Patients randomized to the bosentan 2 mg/kg t.i.d. group who received at least one oral dose of bosentan and who did not violate the protocol in a way that might affect the evaluation of the PK main endpoint.
- Bosentan 2 mg/kg b.i.d. (PK Set): Patients randomized to the bosentan 2 mg/kg b.i.d. group who received at least one oral dose of bosentan and who did not violate the protocol in a way that might affect the evaluation of the PK main endpoint.
Arm/Group | Bosentan 2 mg/kg t.i.d. (PK Set) | Bosentan 2 mg/kg b.i.d. (PK Set)
Number analyzed (Participants) | 27 | 31
h*ng/mL | 7275.1 [5468.2 to 9679.0] | 8535.4 [6936.0 to 10503.7]
Statistical Analysis 1: Comparison: Bosentan 2 mg/kg t.i.d. (PK Set) vs Bosentan 2 mg/kg b.i.d. (PK Set); Test type: Superiority or Other; No statistical test of hypothesis was set for this study. The analysis of PK data was carried out descriptively; Ratio of geometric means = 0.85, 95% CI 2-sided [0.61 to 1.20] — b.i.d. bosentan regimen was taken as reference

2. Other Pre Specified Outcome: Dose-corrected Maximum Plasma Concentration [Cmaxc] of Bosentan
Description: Concentrations of bosentan were measured directly in blood samples collected prior to study drug administration and up to 8 hours or up to 12 hours post-dose for the t.i.d and b.i.d. dosing regimen, respectively.
  The peak plasma concentration (Cmax) of bosentan was directly obtained from the measured plasma concentrations and was dose-corrected to the target dose of 2 mg/kg (Cmaxc).
Time Frame: 0, 0.5, 1, 3, 5 (or 7.5), 8 (or 12 hours) post-dose at Week 4, after at least 2 weeks of stable study drug treatment
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Bosentan 2 mg/kg t.i.d. (PK Set) | Bosentan 2 mg/kg b.i.d. (PK Set)
Number analyzed (Participants) | 27 | 31
ng/mL | 527.9 [386.0 to 721.9] | 742.8 [572.8 to 963.2]
Statistical Analysis 1: Comparison: Bosentan 2 mg/kg t.i.d. (PK Set) vs Bosentan 2 mg/kg b.i.d. (PK Set); Test type: Superiority or Other; No statistical hypothesis tests were set for this study. The analysis of PK data was carried out descriptively; Ratio of geometric means = 0.71, 95% CI 2-sided [0.48 to 1.05] — b.i.d. bosentan regimen was taken as reference

3. Other Pre Specified Outcome: Time to Reach Cmax [Tmax] of Bosentan
Description: Concentrations of bosentan were measured directly in blood samples collected prior to study drug administration and up to 8 hours or up to 12 hours post-dose for the t.i.d and b.i.d. dosing regimen, respectively.
  tmax was obtained directly from the measured plasma concentrations.
Time Frame: 0, 0.5, 1, 3, 5 (or 7.5), 8 (or 12 hours) post-dose at Week 4, after at least 2 weeks of stable study drug treatment
Population: Per protocol PK analysis set (PK set): All patients included in the bosentan 2 mg/kg b.i.d. and bosentan 2 mg/kg t.i.d. groups who received at least one dose of bosentan and who were able to provide at least 5 blood samples for PK assessments and who did not violate the protocol in a way that might affect the evaluation of the PK main endpoint.
Measure: Median (Full Range); unit: hours
Arm/Group | Bosentan 2 mg/kg t.i.d. (PK Set) | Bosentan 2 mg/kg b.i.d. (PK Set)
Number analyzed (Participants) | 27 | 31
hours | 3 [1 to 8] | 3 [0 to 7.5]

4. Other Pre Specified Outcome: Dose-corrected Daily Exposure [AUC(0-24c)] to Bosentan Metabolites (Ro 478634, Ro 485033, Ro 641056)
Description: Concentrations of the metabolites were measured directly in blood samples collected prior to study drug administration and up to 8 hours or up to 12 hours post-dose for the t.i.d and b.i.d. dosing regimen, respectively. Daily exposure to the metabolites corresponds to the area under the concentration-time curve [AUC(0-24)] of the corresponding metabolite over a period of 24 hours, and was calculated in the same manner as the primary endpoint. AUC(0-24c) was corrected to 2 mg/kg (target dose) [AUC(0-24c)].
Time Frame: 0, 0.5, 1, 3, 5 (or 7.5), 8 (or 12 hours) post-dose at Week 4, after at least 2 weeks of stable study drug treatment
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Bosentan 2 mg/kg t.i.d. (PK Set) | Bosentan 2 mg/kg b.i.d. (PK Set)
Number analyzed (Participants) | 27 | 31
h*ng/mL
  AUC(0-24C) for Ro 478634 | 173.2 [126.2 to 237.6] | 200.4 [152.2 to 263.9]
  AUC(0-24C) for Ro 485033 | 968.8 [723.3 to 1297.7] | 1352.5 [1073.4 to 1704.0]
  AUC(0-24C) for Ro 641056 | 716.2 [543.5 to 943.8] | 1014.1 [801.2 to 1283.6]

5. Other Pre Specified Outcome: Change From Baseline in WHO Functional Class at End of Study
Description: The World Health Organization (WHO) defines 4 classes to classify the functional status of patients with pulmonary hypertension (PH):
  Class I (FC I): No limitation of physical activity. Class II (FC II): Slight limitation of physical activity. Class IIII (FC III): Marked limitation of physical activity. Class IV (FC IV): Inability to carry out any physical activity without symptoms.
  Number of patients with improvement (shift from a higher to a lower class), worsening (shift from a lower to a higher class) or no change in WHO functional class at end of study compared to baseline are determined.
Time Frame: Baseline, up to Week 24 on average
Population: All-randomized set. Because all 64 randomized patients were treated with at least one dose of study drug, the All-randomized set was identical to the All-treated set.
Measure: Number; unit: Participants
Groups:
- Bosentan 2 mg/kg t.i.d.: Patients randomized to the bosentan 2 mg/kg t.i.d. group.
- Bosentan 2 mg/kg b.i.d: Patients randomized to the bosentan 2 mg/kg b.i.d. group.
Arm/Group | Bosentan 2 mg/kg t.i.d. | Bosentan 2 mg/kg b.i.d
Number analyzed (Participants) | 31 | 33
Participants
  Worsened WHO FC | 1 | 1
  Unchanged WHO FC | 27 | 25
  Improved WHO FC | 3 | 7

6. Other Pre Specified Outcome: Change From Baseline in Global Clincial Impression Scale (GCIS) at End of Study
Description: The GCIS is an assessment tool providing a single global assessment of the patient's current overall clinical condition: Very Good, Good, Neither Good or Bad, Bad and Very Bad. The assessment was performed both by the physician and the parents / legal representatives independently. Global clinical impression (GCI) at end of study was compared to GCI at baseline and the number of patients with clinical condition considered as worsened, improved or unchanged are determined.
Time Frame: Baseline, up to Week 24 on average
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Bosentan 2 mg/kg t.i.d. | Bosentan 2 mg/kg b.i.d.
Number analyzed (Participants) | 31 | 33
Participants
  Worsened as per physician evaluation | 2 | 2
  Worsened as per parents evaluation | 4 | 3
  Unchanged as per physician evaluation | 24 | 24
  Unchanged as per parents evaluation | 19 | 19
  Improved as per physician evaluation | 5 | 7
  Improved as per parents evaluation | 8 | 11

7. Other Pre Specified Outcome: Number of Patients With Treatment-emergent Liver Function Abnormalities
Description: Number of patients with increase in alanine aminotransferase (ALT) and / or aspartate aminotransferase (AST) above 3 times upper limit of normal (ULN). The worst post-baseline value was considered. The treatment-emergent period was defined as study treatment start date up to 7 calendar days after study treatment end date.
Time Frame: Baseline, up to Week 24
Population: All randomized patients who received at least one dose of study drug and with available data.
Measure: Number; unit: Participants
Groups:
- Bosentan 2 mg/kg t.i.d. (ITT Set): Patients randomized to the bosentan 2 mg/kg t.i.d. group who received at least one oral dose of bosentan.
- Bosentan 2 mg/kg b.i.d. (ITT Set): Patients randomized to the bosentan 2 mg/kg b.i.d. group who received at least one oral dose of bosentan.
Arm/Group | Bosentan 2 mg/kg t.i.d. (ITT Set) | Bosentan 2 mg/kg b.i.d. (ITT Set)
Number analyzed (Participants) | 30 | 33
Participants
  ALT > 3 x ULN | 1 | 0
  AST > 3 x ULN | 0 | 0

8. Other Pre Specified Outcome: Number of Patients With Treatment-emergent Hemoglobin Abnormalities
Description: Number of patients with marked hemoglobin decreases (absolute values below 10 g/dL). The worst post-baseline value was considered.
  The treatment-emergent period was defined as study treatment start date up to 7 calendar days after study treatment end date.
Time Frame: Baseline, up to Week 24
Population: All randomized patients who received at least one dose of study drug and with available data.
Measure: Number; unit: Participants
Arm/Group | Bosentan 2 mg/kg t.i.d. (ITT Set) | Bosentan 2 mg/kg b.i.d. (ITT Set)
Number analyzed (Participants) | 30 | 33
Participants
  Hemoglobin decrease with values < 10 g/dL | 1 | 3
  Hemoglobin decrease with values < 8 g/dL | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study treatment on Day 1 up to 7 days after treatment discontinuation, i.e. up to Week 25 on average
Description: One patient in group 2 mg/kg t.i.d. experienced a serious adverse event (SAE) (adenoviral gastroenteritis) that was reported to the investigator by the parents about 2 months after database closure. Therefore this SAE is not included in the safety summary of FUTURE 3 but is displayed in the cumulative safety data of the FUTURE 3 Extension (AC-052-374)
Groups:
- Bosentan 2 mg/kg t.i.d: Patients received 2 mg/kg of bosentan 3 times a day (morning, afternoon, evening) for at least 0.4 week and up to 28.7 weeks
- Bosentan 2 mg/kg b.i.d: Patients received 2 mg/kg of bosentan twice daily (morning and evening) for at least 6 weeks and up to 26.4 weeks
Arm/Group | Bosentan 2 mg/kg t.i.d | Bosentan 2 mg/kg b.i.d
Serious Adverse Events (participants affected / at risk) | 6/31 | 4/33
Other Adverse Events (participants affected / at risk) | 18/31 | 18/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bosentan 2 mg/kg t.i.d (N=31) | Bosentan 2 mg/kg b.i.d (N=33)
ATRIAL SEPTAL DEFECT REPAIR (Surgical and medical procedures) | 1 (1) | 0 (0)
BODY TEMPERATURE INCREASED (Investigations) | 1 (1) | 0 (0)
BRONCHOPNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (2)
CARDIAC OPERATION (Surgical and medical procedures) | 0 (0) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1)
METABOLIC DISORDER (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
MULTI-ORGAN FAILURE (General disorders) | 0 (0) | 1 (1)
OXYGEN SATURATION DECREASED (Investigations) | 1 (1) | 0 (0)
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PYREXIA (General disorders) | 1 (2) | 0 (0)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1 (1) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bosentan 2 mg/kg t.i.d (N=31) | Bosentan 2 mg/kg b.i.d (N=33)
BRONCHITIS (Infections and infestations) | 1 (1) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 4 (5) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
FLUSHING (Vascular disorders) | 2 (2) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 3 (4) | 5 (8)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 2 (2)
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PYREXIA (General disorders) | 6 (7) | 4 (7)
RASH (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (2) | 2 (3)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 (13) | 6 (8)
VOMITING (Gastrointestinal disorders) | 4 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only agreement between the sponsor and the investigators is that any study-related article or abstract written independently by investigators must be submitted to the sponsor for review at least 60 days prior to submission for publication or presentation.